CLINICAL TRIAL: NCT06933212
Title: Effetto Della DIETa mEdiTerranea Sull'Incidenza di Ictus e Sul Decadimento Cognitivo in Pazienti Affetti da Cadasil e Angiopatia Cerebrale Amiloide
Brief Title: Effect of the Mediterranean Diet in Patients Affected by CADASIL and Cerebral Amyloid Angiopathy.
Acronym: DIETETICA
Status: Recruiting | Type: Observational
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Other Study IDs: DIETETICA
Record Dates: First submitted 2025-04-02; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Cerebral Amyloid Angiopathy; CAA - Cerebral Amyloid Angiopathy
Keywords: CADASIL; CAA; Mediterranean Diet; Nutritional status; Cognitive decline; Stroke incidence
MeSH Terms: conditions — Cerebral Amyloid Angiopathy; Cerebral Amyloid Angiopathy, Familial; CADASIL; Cognitive Dysfunction | interventions — Diet, Mediterranean

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CADASIL
  Interventions: Other: Mediterranean Diet with Extra Virgin Olive Oil; Other: Mediterranean Diet with Walnuts; Other: Low-Fat Control Diet
- CAA patients
  Interventions: Other: Mediterranean Diet with Extra Virgin Olive Oil; Other: Mediterranean Diet with Walnuts; Other: Low-Fat Control Diet

INTERVENTIONS:
Other: Mediterranean Diet with Extra Virgin Olive Oil — participants in this group will follow a Mediterranean Diet enriched with extra virgin olive oil
Other: Mediterranean Diet with Walnuts — participants in this group will follow a Mediterranean Diet enriched with walnuts
Other: Low-Fat Control Diet — participants in this group will follow a low-fat control diet as a comparison to the Mediterranean Diet groups

SUMMARY:
The study is divided into two phases: Phase 1 (observational) and Phase 2 (dietary intervention). The goal of Phase 1 is to assess the nutritional status and dietary habits of two cohorts of patients with CADASIL and CAA. A specific aim is to evaluate adherence to the Mediterranean Diet. The objectives include analyzing patients' nutritional status, lean and fat mass, basal metabolism, and total energy expenditure. It also aims to assess the relationship between adherence to the Mediterranean Diet and the onset of stroke and cognitive decline, as well as examine stroke severity (ischemic or hemorrhagic) and its association with Mediterranean Diet adherence (MEDAS questionnaire). Additionally, the study will explore the link between diet adherence and cognitive deficits, and measure changes in biological and anthropometric parameters as a result of adopting the Mediterranean Diet.

Phase 2 is an interventional dietary study designed to evaluate the effects of the Mediterranean Diet, enriched with either extra virgin olive oil or walnuts, on stroke incidence and cognitive decline in patients with CAA and CADASIL.

ELIGIBILITY:
Inclusion Criteria:

* The study will include individuals of both sexes aged 18 years or older with a diagnosis of CADASIL (confirmed genetically by the presence of the NOTCH3 gene mutation) or possible/probable CAA (defined according to the Boston 2.0 criteria). All participants must provide informed consent for the use of demographic, clinical, and nutritional data for scientific purposes in an anonymous form

Exclusion Criteria:

* na

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with CADASIL and CAA who are referred to the outpatient clinics and hospital department of the Complex Structure "Neurology 9 - Cerebrovascular Diseases" at the Fondazione IRCCS Istituto Neurologico "Carlo Besta" in Milan will be enrolled in the study. All patients will be asked to provide their consent to participate in the study by signing a specific form that includes consent for the collection of demographic, clinical, and nutritional data.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Stroke | Throughout the study, from baseline to the end of the study (12 months or as specified).
  evaluation of the incidence of stroke (ischemic and hemorrhagic) in patients following the Mediterranean Diet (with olive oil or walnuts) compared to a low-fat control diet. The incidence of stroke (ischemic and hemorrhagic) will be assessed through clinical diagnosis, based on medical records and confirmed by neuroimaging techniques (e.g., MRI, CT scans). Stroke type (ischemic or hemorrhagic) will be classified based on neuroimaging results and clinical evaluation.
Cognitive Decline | Throughout the study, from baseline to the end of the study (12 months or as specified).
  Cognitive decline will be assessed using the Montreal Cognitive Assessment (MoCA), a standardized neuropsychological test. The MoCA scale ranges from 0 to 30, with higher scores indicating better cognitive function and lower scores suggesting greater cognitive impairment. The MoCA score is corrected for the patient's age and education level. A corrected score below 18.59 indicates cognitive impairment below the normal range. A score between 18.59 and 20.69 suggests the patient is within the lower limits of the normal range, while a score above 20.69 indicates a score above the normal range, according to Italian reference norms. The test will be administered by a trained neuropsychologist

SECONDARY OUTCOMES:
Adherence to Mediterranean Diet | Baseline, 6 months, and 12 months
  Adherence to Mediterranean Diet is assessed using Mediterranean Diet Adherence Screener (MEDAS), a validated 14-item questionnaire. A total MEDAS score is calculated by summing the points from all items, obtaining a score ranging from 0 to 14. Subjects with scores above 9 are classified as having high adherence to the MD, those scoring between 6 and 8 have moderate adherence, and scores below 6 indicate low adherence.
Nutritional Status | Baseline and 12 months.
  Physical activity level is assessed using the validated 7-item International Physical Activity Questionnaire (IPAQ), which evaluates activity over the past 7 days. Activity volume is calculated by weighting each activity type according to its energy expenditure, expressed in metabolic equivalents (METs), and the total daily METs for each patient is determined. Mini Nutritional Assessment (MNA) is used to identify malnourished patients or those at risk of malnutrition in elderly individuals in clinics, hospitals and nursing homes. MNA is a validated test of 18 multiple choice questions divided into two parts. A final score which indicates the level of the risk of malnutrition (low, medium or high), is obtained. A score between 24-30 indicates an adequate nutritional status, 17-23.5 shows a risk of malnutrition and a value < 17 is an indicator of malnutrition or poor nutritional status
Body Composition (Lean and Fat Mass) | Baseline and 12 months.
  Anthropometric measurements are collected according to the conventional criteria and measuring procedures proposed by Lohman. All patients undergo the following anthropometrics measurements: body weight (kg), body height (cm), body circumference (cm) and skinfold thickness (mm). Each skinfold thickness is measured 3 times and the mean value is calculated. Body density and fat mass are calculated using the Durnin and Womersley method and by Siri formula, respectively. Fat mass is then converted to kilograms, which allows for the estimation of fat-free mass in kilograms. All the measurements are performed on the non-dominant side of the body
Basal Metabolism and Total Energy Expenditure | Baseline and 12 months.
  Through METs calculations, the physical activity level is estimated, enabling the estimation of total daily energy expenditure (TDEE) using the basal metabolic rate (BMR) determined by Harris-Benedict formula.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tuttolomondo A, Di Raimondo D, Casuccio A, Velardo M, Salamone G, Arnao V, Pecoraro R, Della Corte V, Restivo V, Corpora F, Maida C, Simonetta I, Cirrincione A, Vassallo V, Pinto A. Relationship between adherence to the Mediterranean Diet, intracerebral hemorrhage, and its location. Nutr Metab Cardiovasc Dis. 2019 Oct;29(10):1118-1125. doi: 10.1016/j.numecd.2019.06.010. Epub 2019 Jun 20. PMID 31383501
- [Background] Tuttolomondo A, Simonetta I, Daidone M, Mogavero A, Ortello A, Pinto A. Metabolic and Vascular Effect of the Mediterranean Diet. Int J Mol Sci. 2019 Sep 23;20(19):4716. doi: 10.3390/ijms20194716. PMID 31547615
- [Background] Misirli G, Benetou V, Lagiou P, Bamia C, Trichopoulos D, Trichopoulou A. Relation of the traditional Mediterranean diet to cerebrovascular disease in a Mediterranean population. Am J Epidemiol. 2012 Dec 15;176(12):1185-92. doi: 10.1093/aje/kws205. Epub 2012 Nov 27. PMID 23186748
- [Background] Tuttolomondo A, Casuccio A, Butta C, Pecoraro R, Di Raimondo D, Della Corte V, Arnao V, Clemente G, Maida C, Simonetta I, Miceli G, Lucifora B, Cirrincione A, Di Bona D, Corpora F, Maugeri R, Iacopino DG, Pinto A. Mediterranean Diet in patients with acute ischemic stroke: Relationships between Mediterranean Diet score, diagnostic subtype, and stroke severity index. Atherosclerosis. 2015 Nov;243(1):260-7. doi: 10.1016/j.atherosclerosis.2015.09.017. Epub 2015 Sep 11. PMID 26409625
- [Background] Feart C, Samieri C, Alles B, Barberger-Gateau P. Potential benefits of adherence to the Mediterranean diet on cognitive health. Proc Nutr Soc. 2013 Feb;72(1):140-52. doi: 10.1017/S0029665112002959. Epub 2012 Dec 11. PMID 23228285
- [Background] Shannon OM, Ranson JM, Gregory S, Macpherson H, Milte C, Lentjes M, Mulligan A, McEvoy C, Griffiths A, Matu J, Hill TR, Adamson A, Siervo M, Minihane AM, Muniz-Tererra G, Ritchie C, Mathers JC, Llewellyn DJ, Stevenson E. Mediterranean diet adherence is associated with lower dementia risk, independent of genetic predisposition: findings from the UK Biobank prospective cohort study. BMC Med. 2023 Mar 14;21(1):81. doi: 10.1186/s12916-023-02772-3. PMID 36915130
- [Background] Roman GC, Jackson RE, Gadhia R, Roman AN, Reis J. Mediterranean diet: The role of long-chain omega-3 fatty acids in fish; polyphenols in fruits, vegetables, cereals, coffee, tea, cacao and wine; probiotics and vitamins in prevention of stroke, age-related cognitive decline, and Alzheimer disease. Rev Neurol (Paris). 2019 Dec;175(10):724-741. doi: 10.1016/j.neurol.2019.08.005. Epub 2019 Sep 11. PMID 31521398
- [Background] Lin B, Hasegawa Y, Takane K, Koibuchi N, Cao C, Kim-Mitsuyama S. High-Fat-Diet Intake Enhances Cerebral Amyloid Angiopathy and Cognitive Impairment in a Mouse Model of Alzheimer's Disease, Independently of Metabolic Disorders. J Am Heart Assoc. 2016 Jun 13;5(6):e003154. doi: 10.1161/JAHA.115.003154. PMID 27412896
- [Background] Biffi A, Greenberg SM. Cerebral amyloid angiopathy: a systematic review. J Clin Neurol. 2011 Mar;7(1):1-9. doi: 10.3988/jcn.2011.7.1.1. Epub 2011 Mar 31. PMID 21519520
- [Background] Buffon F, Porcher R, Hernandez K, Kurtz A, Pointeau S, Vahedi K, Bousser MG, Chabriat H. Cognitive profile in CADASIL. J Neurol Neurosurg Psychiatry. 2006 Feb;77(2):175-80. doi: 10.1136/jnnp.2005.068726. PMID 16421118
- [Background] Ruchoux MM, Maurage CA. CADASIL: Cerebral autosomal dominant arteriopathy with subcortical infarcts and leukoencephalopathy. J Neuropathol Exp Neurol. 1997 Sep;56(9):947-64. PMID 9291937
- [Background] Chabriat H, Joutel A, Dichgans M, Tournier-Lasserve E, Bousser MG. Cadasil. Lancet Neurol. 2009 Jul;8(7):643-53. doi: 10.1016/S1474-4422(09)70127-9. PMID 19539236